CLINICAL TRIAL: NCT02269566
Title: A Double-blinded Placebo-controlled Randomized Clinical Trial Evaluating the Efficacy and Adverse Effect of Intralymphatic Immunotherapy (ILIT) for House Dust Mite, Cat, and Dog Allergen in Allergic Rhinitis Patients
Brief Title: Intralymphatic Immunotherapy (ILIT) for House Dust Mite, Cat, and Dog Allergen in Allergic Rhinitis Patients
Acronym: ILIT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The number of enrolled subjects did not meet the goal during the study
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Principal Investigator, Sang Min Lee, Assistant professor of Division of Pulmonology and Allergy, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140101480
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allergen extract (Active Comparator): 0.1 ml of allergen extracts
  Interventions: Drug: HollisterStier
- Placebo (Placebo Comparator): Normal saline, 0.1 ml
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: HollisterStier — 0.1 ml of 30 AU/ml for Df or Dp, 10 AU/ml for Cat hair, and/or 1:1/10 weight/volume for dog hair/dander 3 injections into an inguinal lymph node
  Other Names: Allergen extracts, New Orleans, USA
  Arms: Allergen extract
Drug: Normal saline — 0.1 ml of normal saline 3 injections into an inguinal lymph node
  Other Names: JW-pharma, Seoul, Republic of Korea
  Arms: Placebo

SUMMARY:
We will perform double-blinded placebo-controlled randomized clinical trial which evaluates the efficacy and safety of allergen-specific intralymphatic immunotherapy (ILIT) for allergens including Dermatophagoides farinae (Df), Dermatophagoides pteronyssinus (Dp), cat, and dog that are sensitized and provoke rhinitis-related symptoms in patients with allergic rhinitis.

DETAILED DESCRIPTION:
After informed consent, subjects will be randomly assigned to ILIT group or placebo group in double-blind manner. In both group, causal allergen or placebo will be injected into inguinal lymph node through guidance by ultrasonography three times with 4-week interval. In ILIT group, initial dose of allergen will be 1,000-fold diluted solution from maximal concentration of allergen extract for subcutaneous immunotherapy (30 AU/ml for Df or Dp, 10 AU/ml for Cat hair, and 1:1/10 weight/volume for dog hair/dander, HollisterStier, New Orleans, USA) in volume of 0.1ml. If skin is highly reactive in skin prick test, the initial dose will be 10-fold dilution from maximal concentration where diameter of wheal is less than that of histamine. After the first dose, allergen concentration will be escalated 3-fold at second dose, and 10-fold at third dose if there are no local or systemic hypersensitivity reaction. The allergen concentration will not change at second or third dose if there is mild local or systemic reaction. The allergen concentration will decrease by 10 or 100-fold from previous concentration or further injection will be holded if there is severe local or systemic reaction after sufficient explanation and discussion with subjects.

The investigators will evaluate allergic rhinitis symptom score before and 4, 12 months after the initial treatment. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) and Sino-Nasal Outcome Test (SNOT-20) will be used. Visual analogue scale (VAS) of symptoms including rhinorrhea, sneezing, nasal obstruction, postnasal drip, eye/nose/ear/palate itching, dyspnea, wheezing, chest discomfort as well as urticaria, angioedema, and itching on exposed skin during exposure to causal allergen in daily life will be also evaluated. Skin prick test, intradermal test, blood sampling for serum allergen-specific IgE, exhaled nitric oxide, and nasal lavage for Th1, Th2, and Treg cytokines will be also performed before and 4, 12 months after the initial treatment.

Adverse events will be recorded and graded according to Muller classification and Ring and Messner classification.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis to house dust mite (Df, Dp), cat or dog
* More than 3mm reaction at skin prick test for Df, Dp, cat or dog or more than class 3 at serum specific IgE level (UNICAP or MAST)

Exclusion Criteria:

* Uncontrolled or severe asthma according to Global Initiative of Asthma (GINA) guideline
* FEV1 less than 50% of predicted value if there is comorbid asthma.
* Subject rejects the enrollment into study
* Low compliance
* Pregnancy or lactation
* Significant cardiovascular, hepatic, renal, hematologic, oncologic, or infectious diseases
* Administration of beta blocker, angiotensin converting enzyme inhibitor, tricyclic antidepressant, immnosuppressant including systemic glucocorticosteroid (20mg or more dose of prednisolone or equivalent dose of other steroid) within last 2 weeks
* Prior history of allergen-specific immunotherapy
* Allergic rhinitis caused by other perennial or seasonal allergen
* Vulnerable volunteer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire | up to 12 months after the initial treatment

SECONDARY OUTCOMES:
SNOT-20 | before and 4, 12 months after the initial treatment
  Sino-Nasal Outcome Test
Skin reactivity | before and 4, 12 months after the initial treatment
  Diameters of wheal provoked by causal allergens in skin prick test and intradermal test
Serum alllergen-specific IgE level | before and 4, 12 months after the initial treatment
  Serum alllergen-specific IgE level using UNICAP, Thermofisher Scientific, Sweden
Nasal reactivity | before and 4, 12 months after the initial treatment
  Threshold concentration in nasal provocation test for allergens of Df and Dp
Cytokines in nasal lavage fluid | before and 4, 12 months after the initial treatment
  Cytokines of Th1, Th2, and Treg in nasal lavage fluid
Exhaled NO | before and 4, 12 months after the initial treatment
  Exhaled nitric oxide measuring NIOX MINO, Thermofisher Scientific, Sweden
Allergic rhinitis symptoms during allergen exposure in daily life | before and 4, 12 months after the initial treatment
  Visual analog scare of allergic rhinitis symptoms during allergen exposure in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, M.D., Ph.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Background] Martinez-Gomez JM, Johansen P, Erdmann I, Senti G, Crameri R, Kundig TM. Intralymphatic injections as a new administration route for allergen-specific immunotherapy. Int Arch Allergy Immunol. 2009;150(1):59-65. doi: 10.1159/000210381. Epub 2009 Apr 2. PMID 19339803
- [Background] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy. Curr Opin Allergy Clin Immunol. 2009 Dec;9(6):537-43. doi: 10.1097/ACI.0b013e3283310ff7. PMID 19680119
- [Background] von Moos S, Kundig TM, Senti G. Novel administration routes for allergen-specific immunotherapy: a review of intralymphatic and epicutaneous allergen-specific immunotherapy. Immunol Allergy Clin North Am. 2011 May;31(2):391-406, xi. doi: 10.1016/j.iac.2011.02.012. PMID 21530827
- [Background] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Background] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Background] Witten M, Malling HJ, Blom L, Poulsen BC, Poulsen LK. Is intralymphatic immunotherapy ready for clinical use in patients with grass pollen allergy? J Allergy Clin Immunol. 2013 Nov;132(5):1248-1252.e5. doi: 10.1016/j.jaci.2013.07.033. Epub 2013 Sep 13. No abstract available. PMID 24035151
- [Background] Kundig TM, Johansen P, Bachmann MF, Cardell LO, Senti G. Intralymphatic immunotherapy: time interval between injections is essential. J Allergy Clin Immunol. 2014 Mar;133(3):930-1. doi: 10.1016/j.jaci.2013.11.036. Epub 2014 Jan 15. No abstract available. PMID 24439076
- [Background] Zaleska A, Eiwegger T, Soyer O, van de Veen W, Rhyner C, Soyka MB, Bekpen C, Demiroz D, Treis A, Sollner S, Palomares O, Kwok WW, Rose H, Senti G, Kundig TM, Ozoren N, Jutel M, Akdis CA, Crameri R, Akdis M. Immune regulation by intralymphatic immunotherapy with modular allergen translocation MAT vaccine. Allergy. 2014 Sep;69(9):1162-70. doi: 10.1111/all.12461. Epub 2014 Jul 12. PMID 24934402